CLINICAL TRIAL: NCT04637984
Title: The Implementation of PREP2 Algorithms Into Clinical Practice: a Strategy for Improving Rehabilitation Efficiency and Clinical Outcomes After Stroke. A Single-site Randomized Control Trial
Brief Title: The Implementation of PREP2 Algorithm Into Clinical Practice
Acronym: PRESTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Sofia Straudi, Clinical Professor, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Predict_stroke_outcomes
Record Dates: First submitted 2020-10-29; First posted 2020-11-20 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Rehabilitation
Keywords: rehabilitation efficiency; PRESTO algorithms; physical rehabilitation; stroke; motion kinematics; brain activity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Implementation Group (Experimental): Predictions will be provided to the rehabilitation team and discussed with the patient and their family. Patients will receive a multidisciplinary rehabilitation according to their individual needs.
  Interventions: Behavioral: PREP2 algorithm
- Control Group (No Intervention): This group will not received any information on the PREP2

INTERVENTIONS:
Behavioral: PREP2 algorithm — A) PREP2. It combines clinical measures and neurological biomarkers in the initial days after stroke: 1) SAFE score (day 3), which is the sum of shoulder abduction and finger extension strength in the paretic upper limb using the Medical Research Council (MRC); 2) NIH Stroke Scale (day 3); 3) transcranial magnetic stimulation (day 3-7) to determine the presence of MEPs in the paretic arm. According with the aforementioned measures, 4 categories of upper limb recovery will be identified: EXCELLENT, GOOD, LIMITED and POOR.
  Arms: Implementation Group

SUMMARY:
Stroke is a worldwide major cause of disability with great social and economic burdens. The recovery of motor function is crucial for the patient to regain independence and quality of life. Identifying early predictors of motor recovery and outcomes is useful for planning personalized rehabilitation programs and increasing their efficiency. However, making predictions using a single clinical assessment is often difficult and a combination of multiple tools is required. In the last decades, were validated two predictive algorithms for upper limb function and independent walking that can be easily implemented into clinical practice with the aim of increasing knowledge on expected outcome after stroke in patients, families and rehabilitation teams. This will be the first single-site randomized control trial that will test the implementation of such tools in a rehabilitation setting in Italy.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of stroke;
* new upper and/or lower limb weakness.

Exclusion Criteria:

* cerebellar or bilateral stroke;
* contraindication to TMS;
* cognitive or communication impairment precluding informed consent;
* assisted walking prior to admission;
* severe medical conditions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Rehabilitation LOS (days) | Hospital discharge (an average of 3-6 months)
  Length of stay as measure of rehabilitation efficiency
Change in Functional International Measure between two time points | Baseline, hospital discharge (an average of 3-6 months)
  Measure of efficiency of rehabilitation. Assess a patient's level of disability as well as change in patient status in response to rehabilitation.
Change in Rehabilitation Complexity Scale between two time points | Baseline, hospital discharge (an average of 3-6 months)
  Measure of the complexity of rehabilitation needs and/or interventions.
Change in Rehabilitation strategies between two time points | Baseline, week 4
  Will be assessed tracking: therapists confidence about patients' recovery (0-5 Likert scale); therapy content; therapy duration.
Change in Action Research Arm Test between three time points | week 4, 12, week 26
  To assess upper extremity performance (coordination, dexterity and functioning)
Change in Fugl-Meyer Assessment between three time points | week 4, 12, week 26
  To assess the sensorimotor impairment in individuals who have had stroke.
Change in Stroke Impact Scale 3.0 between three time points | week 4, 12, week 26
  To evaluate how stroke has impacted your health and life.
Change in Electroencephalography power in beta band between three time points | week 4, week 12, week 26
  EEG data will be recorded with the aim of characterizing the PREP2 recovery classes.
Change in Electroencephalography power in alpha band between three time points | week 4, week 12, week 26
  EEG data will be recorded with the aim of characterizing the PREP2 recovery classes.
Change in Kinematic data recordings between three time points | week 4, week 12, week 26
  Kinematic data of trunk and affected hand will be recorded during subject imitations. Kinematic data will be recorded with the aim of characterizing the PREP2 recovery classes.

SECONDARY OUTCOMES:
Applicability perception and satisfaction degree of the proposed intervention self-report questionnaire. | week 4
  Self-report questionnaire using a Visual Analogue Scale (0 - Strongly disagree; 10 - Strongly agree). Higher score indicates greater satisfaction with the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neuroscience and Rehabilitation, University Hospital of Ferrara, Ferrara, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: Undecided